CLINICAL TRIAL: NCT03463603
Title: Ethnic Differences in Acute Coronary Syndromes Care in Emergency Departments.
Acronym: ASCEND
Status: Completed | Type: Observational
Sponsor: University of British Columbia (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government); Michael Smith Foundation for Health Research (Other); Heart and Stroke Foundation of Canada (Other)
Responsible Party: Principal Investigator, Martha Mackay, Clinical Associate Professor, University of British Columbia
Other Study IDs: H13-00617
Record Dates: First submitted 2018-02-05; First posted 2018-03-13 (Actual); Last update posted 2018-03-14 (Actual); Status verified 2018-03

CONDITIONS: Acute Coronary Syndrome; Racial Bias
Keywords: ischemic heart disease; acute coronary syndrome; racial bias
MeSH Terms: conditions — Acute Coronary Syndrome; Racism; Myocardial Ischemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Asian racial identity: Those who self-report "Asian" or related terms as their racial identity.
- South Asian racial identity: Those who self-report "South Asian" or related terms as their racial identity.
- Other racial identity: All others, who self-report neither "Asian", "South Asian" or their related terms as their racial identity.

SUMMARY:
When doctors and nurses use accepted guidelines for quickly treating patients who come to the emergency department (ED) with a possible heart attack, patients do better. Research shows that there are racial-identity- and ethnicity-based differences in the symptoms these patients have, when and why they seek care, the treatments they receive, and how well they fare afterwards. There is also Canadian evidence that there may be racial-identity-based disparities in the care some patients receive, and it has been suggested that health professionals may unconsciously treat patients of different racial identities differently. But it is not known if there is racial-identity variation in the care given to Canadian patients with heart attack symptoms in the critical first hours after coming to an ED, or in their experiences of this care. The investigators collected information from the health records of patients who come to EDs with symptoms of heart attack. The investigators recorded events and times such as what provisional diagnosis was assigned to the patient, how often they received pain medication, how long until certain tests were performed and what treatments were offered. The investigators also collected information about things that might affect delivery of care, e.g., the number of doctors and nurses who were on duty. Participants also completed a short questionnaire about their reasons for coming to the hospital, how long they waited before coming and why, and what their experience in the ED was like. The investigators reviewed this information to see if there are racial-identity-based differences in the care received by patients with heart attack symptoms. The findings could identify important disparities, which could in turn inform future projects to correct these disparities, for example, education of health professionals about ethnic differences in ideas of health and illness.

DETAILED DESCRIPTION:
The investigators conducted a prospective, observational study in which patients presenting to EDs who were subsequently diagnosed with acute coronary syndrome (ACS) or possible ACS were identified. The investigators collected data related to receiving the accepted standard of care for ACS patients. Information about the participants' initial symptoms, attribution of their symptoms, treatment-seeking choices, and perceptions of the care received in the ED was collected.

Setting and Sample: The investigators conducted the study at three sites: Hospital 1 is in an inner-city, quaternary care, university-affiliated hospital whose ED has approximately 71,000 patient visits annually, about 2,800 of which are patients with symptoms that are potentially due to myocardial ischemia. The medical and nursing staffing levels are staggered based on expected patient volumes, ranging from 15 to 18 registered nurses (RNs) and 1 to 6 physicians at a given time. There are also support staff, including licensed practical nurses, aides; clerks, ECG technicians, etc. There is a designated triage area, staffed continuously by at least one RN. Hospital 2's ED is in a large community hospital in a different health authority. It has 100,000 patient visits annually, approximately 6,500 of which are patients with potentially ischemic symptoms. The medical and nursing staffing levels are similar to the first site, ranging from 19 to 22 registered nurses (RNs) and 1 to 4 physicians at a given time. This site is in a community with a very high proportion of South Asian people (27.5%). Hospital 3 is also a community hospital with fewer ED visits annually, but similar nursing and medical staffing levels. This site is in a community with a very high proportion (52.5%) of people identifying as being of Chinese ancestry.

Procedures: Research assistants (RAs) fluent in English, Mandarin and Cantonese for the tertiary site and one fluent in English and Punjabi for the community site recruited participants.

Recruitment. The RAs identified potential participants, seven days per week, from one of three sources: (1) a list, obtained daily from the ED charge nurse, of all patients admitted to the hospital since the RA's last visit who were triaged with codes related to a possible ACS; (2) the current charge nurse, who identified any patient currently in the ED who met study criteria as signified by the ED physician ordering one of the following: (i) cardiology consult, (ii) cardiac computational tomography, or (iii) 2- or 6-hour repeat cardiac biomarker and ECG, followed by outpatient provocative stress testing; (3) a list, obtained from the stress-testing laboratory, of all patients who had been referred from the ED for urgent (within 48 hours) outpatient stress testing.

Recruitment occurred in the ED, the cardiology units (CCU or telemetry unit) and in the stress-testing laboratory. Potential participants were screened for general eligibility through discussion with the nurse or cardiology technologist. Those believed to be eligible were approached and invited to participate.

Data collection. Data regarding delivery of guideline-based care in the ED were collected from the health record (e.g., time to stretcher, time to ECG, time to first MD assessment, medications administered) and other processes (e.g., occurrence and timing of cardiology consultation, transfer from ED to a critical care area). Data regarding several patient-, environment- and system-related potential covariates were collected from the health record (e.g., mode of arrival at ED; language spoken; accompanied by family/friend; language ability of family/friend; symptoms reported) and ED staffing records (staffing levels). Data pertaining to the entire ED stay were captured.

Participants were asked to respond to a questionnaire, administered by the RA, regarding their decision to seek treatment and their perspectives on their ED care. Ethnicity, racial identity and other sociodemographic data were obtained during the interview.

For those admitted to the hospital, additional data regarding admission unit , procedures offered, refused and undergone, major adverse cardiac events, length of stay and final diagnosis were collected. For participants who were discharged from the ED with referral to outpatient stress testing, we tracked discharge diagnosis, attendance at, and interpretation of the test.

Measures: The primary outcome variable, door-to-ECG time, was defined as the time from triage to first ECG acquisition. The official triage time is the time entered by the triage nurse when the patient is initially evaluated. The time of the first ECG is an electronic time stamp appearing in the clinical information system, entered when the ECG is acquired.

The predictor variables ethnicity and racial identity were measured by self-report.

Other outcome variables and potential confounders:

1. Time intervals: Several time intervals were measured, based on the official triage time.
2. Location, nature and severity of reported symptoms: All symptoms reported by participant, as well as their intensity.
3. Acuity at time of triage: measured using the Canadian Triage and Acuity Score. The participants' presenting complaint was measured using the Canadian Emergency Department Information System standardised codes, in use at the study sites.
4. Other data: Mode of transport to hospital, accompanied versus alone, noted difficulty with English, presence of interpreter during care
5. Number and frequency of physician and nurse assessments/interventions.
6. Measured clinical parameters: All documented observations of ECG rhythm and vital signs.
7. Medications: Agent, dose, route and time of administration
8. Diagnostic testing: Timing and frequency of bloodwork and ECGs.
9. Consultation: Consultation of other medical services.
10. Patient Disposition.
11. Patient perspectives: Time of onset, type of symptoms, decisions to seek treatment and reasons for delaying; participants' perspectives on care in ED; other socio-demographic variables
12. Emergency department contextual factors: Staffing levels for each shift.
13. Post-ED care: Diagnostic tests and interventions offered and completed after leaving ED, e.g., referral for / offer of / consent to / receipt of angiogram, percutaneous coronary intervention or cardiac surgery; discharge diagnosis; length of hospital stay.

ELIGIBILITY:
Inclusion Criteria:

* 20 years of age or older
* presented to the ED and are either referred for immediate cardiology consultation or managed according to a standardized protocol for continued observation and referral for follow-up (whether ultimately admitted or not);
* hemodynamically stable and free of ischemic discomfort for at least one hour
* spoke English, Mandarin, Cantonese, Punjabi
* able to provide informed consent.

Exclusion Criteria:

• being cared for by any of the Emergency physicians (3) who were co-investigators

Min Age: 20 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients presenting to Emergency Departments with symptoms suggestive of an acute coronary syndrome.
Sampling Method: Non-Probability Sample
Enrollment: 448 (Actual)
Dates: Start 2013-10-07 (Actual); Primary Completion 2017-01-11 (Actual); Study Completion 2017-04-12 (Actual)

PRIMARY OUTCOMES:
Door to ECG | from hour and minute of admission until the hour and minute of first documented ECG, up to 48 hours
  time from Emergency triage to first ECG acquisition

SECONDARY OUTCOMES:
Number of assessments by health professionals | from hour and minute of admission until the hour and minute of transfer to inpatient unit or discharge from Emergency Department, whichever comes first, up to 48 hours
  The number of assessments by physicians and nurses during the ED stay.
Rate of being offered and consenting to coronary angiogram | from date of admission until the date of hospital discharge, up to 100 weeks
  Rate of being offered and consenting to coronary angiogram among those having a diagnosis of acute coronary syndrome or myocardial infarction.
Rate of being offered and consenting to any revascularization procedure | from date of admission until the date of hospital discharge, up to 24 weeks
  Rate of being offered and consenting to any revascularization procedure among those having coronary atherosclerotic lesions >/= 70% in any vessel
ethnic differences in treatment-seeking delay | from hour and minute of first documented symptoms until the hour and minute of first documented help-seeking, up to 168 hours
  the time between symptom onset and the decision to seek medical help

CONTACTS AND LOCATIONS:
Locations (3):
- Canada (3):
  - Richmond Hospital, Richmond, British Columbia
  - Surrey Memorial Hospital, Surrey, British Columbia
  - St. Paul's Hospital, Vancouver, British Columbia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Iacoe E, Ratner PA, Wong ST, Mackay MH. A cross-sectional study of ethnicity-based differences in treatment seeking for symptoms of acute coronary syndrome. Eur J Cardiovasc Nurs. 2018 Apr;17(4):297-304. doi: 10.1177/1474515117741893. Epub 2017 Nov 15. PMID 29140107
- [Result] Mackay, M.H., Ratner, P.A., Scheuermeyer, F.X., Veenstra, G., Ramanathan, K.R., O'Sullivan, M.E., Grubisic, M., Murray, C., Humphries, K.H. (2017). Is racism a factor in emergency department care of patients with suspected acute coronary syndrome? Canadian Journal of Cardiology, 33 (10), s125-126.